CLINICAL TRIAL: NCT00749320
Title: Arterial Spin Labeling Blood Flow Magnetic Resonance Imaging for the Evaluation of Response to Antiangiogenic and Targeted Therapies of Metastatic Renal Cell Carcinoma
Brief Title: Arterial Spin Labeling Blood Flow MRI for Evaluation of Response to Antiangiogenic and Targeted Therapies of Renal Cell Carcinoma (RCC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); Pfizer (Industry); Novartis (Industry)
Responsible Party: Principal Investigator, Leo Tsai, MD, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 08-078
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Renal Cell Carcinoma
Keywords: MRI; Sunitinib; Pazopanib
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ASL MRI (Other): ASL MRI performed at different time intervals on participants receiving sunitnib or pazopanib for treating RCC
  Interventions: Other: Arterial Spin Labeling Magnetic Resonance Imaging

INTERVENTIONS:
Other: Arterial Spin Labeling Magnetic Resonance Imaging — ASL MRI performed at different time intervals on participants receiving sunitinib or pazopanib for treating RCC
  Other Names: ASL MRI

SUMMARY:
The purpose of this study is to assess magnetic resonance imaging (MRI) as a tool to track tumor growth for renal cell carcinoma while the participant is receiving clinical treatment therapy with sunitinib or pazopanib. An MRI is a sophisticated type of scan that uses powerful magnets to make clearer images or to focus on detailed medical information in the participants abdomen and pelvis. This imaging done for this study will use the ASL MRI technique that allows us to see blood flow changes which possibly may indicated tumor growth.

DETAILED DESCRIPTION:
* MRI's will be performed at specific time points during the participants treatment for renal cell carcinoma with the drug sunitinib or pazopanib. These ASL MRI's will be performed at baseline, 2 weeks upon initiation of therapy with sunitinib/pazopanib, after cycle 2 and/or cycle 4 of therapy, and at the end of therapy.
* The MRI tests for all participants will be done at Beth Israel Deaconess Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with metastatic renal cell carcinoma and who will initiate sunitinib or pazopanib
* Enrolled on protocol 06-105, "Collection of specimens and clinical data from patients with renal cell carcinoma treated with targeted therapies," or receiving Pazopanib as part of routine clinical care.
* Found to have tumors that are 2.5cm or greater as determined by CT imaging
* Candidate lesions for ASL MRI should be 2.5cm or greater. Order of preference of lesion location will be as follows: abdominal lesions, bone lesions and chest lesions

Exclusion Criteria:

* Contraindication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-09; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
To explore the association of baseline blood flow in renal cell carcinoma measured by ASL MRI and tumor response to treatment with sunitinib or pazopanib | 2 years
To explore the association of changes in tumor blood flow that occur early in the course of therapy compared to baseline and response of RCC to treatment with sunitinib or pazopanib | 2 years
To evaluate the association between canges in tumor blood flow on ASL over the course of therapy and at the time of disease progression and resistance to therapy | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Leo Tsai, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Derived] Tsai LL, Bhatt RS, Strob MF, Jegede OA, Sun MRM, Alsop DC, Catalano P, McDermott D, Robson PM, Atkins MB, Pedrosa I. Arterial Spin Labeled Perfusion MRI for the Evaluation of Response to Tyrosine Kinase Inhibition Therapy in Metastatic Renal Cell Carcinoma. Radiology. 2021 Feb;298(2):332-340. doi: 10.1148/radiol.2020201763. Epub 2020 Dec 1. PMID 33258745